CLINICAL TRIAL: NCT06341972
Title: Improving Psychological Outcomes for Acute Respiratory Failure Survivors Using a Self-Management Intervention
Acronym: SMARA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Francis Family Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00247005; K23HL155735 (NIH)
Record Dates: First submitted 2024-03-25; First posted 2024-04-02 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Failure; Anxiety; Critical Illness
MeSH Terms: conditions — Respiratory Insufficiency; Anxiety Disorders; Critical Illness

STUDY DESIGN:
Intervention Model Description: pilot randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-management intervention (Experimental): Cognitive behavioral therapy based self-management intervention for anxiety
  Interventions: Behavioral: Cognitive behavioral therapy based self-management for anxiety
- Usual Care (No Intervention): Usual hospital-based care

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy based self-management for anxiety — Evidenced based approach for educating patients about how to manage anxiety after respiratory failure.
  Other Names: SMARA
  Arms: Self-management intervention

SUMMARY:
A growing number of patients are surviving a stay in the intensive care unit (ICU) but may experience long-lasting psychological problems, but research evaluating such treatment for ICU patients is scant.

The goal of this pilot randomized controlled trial is to evaluate the feasibility, acceptability, and potential benefit of an evidence-based psychological intervention for anxiety and associated outcomes for ICU patients.

The main question[s] it aims to answer are:

* Is this intervention feasible and acceptable in ARF patients?
* Is this intervention in the ICU and hospital associated with reduced anxiety symptoms?

Participants will participate in a cognitive behavioral therapy informed self-management intervention aimed to reduce anxiety symptoms. Researchers will compare the intervention group to patients who receive usual care to see if the intervention reduces symptoms at the the conclusion of the intervention and at 3 months follow-up.

DETAILED DESCRIPTION:
Statement of the Problem. An increasing number of adults develop acute respiratory failure (ARF) requiring mechanical ventilation in an intensive care unit (ICU). To improve patient outcomes, evidence-based guidelines recommend titrating sedatives to allow for patient wakefulness while in the ICU. However, among awake acute respiratory failure patients, anxiety can be a common and long-lasting problem. Outside of the ICU setting, cognitive behavioral therapy based self-management is an established, evidence-based, first-line treatment for patients with anxiety. However, there is limited evidence about the feasibility and benefit of cognitive behavioral therapy interventions for acute respiratory failure patients with anxiety during hospitalization.

Specific Aims. This award proposal seeks to conduct a pilot randomized controlled trial of a tailored self-management protocol vs. usual care in the ICU and subsequent hospital ward to establish its feasibility, acceptability (primary outcome; Aim 1a), and potential efficacy in reducing anxiety symptoms and associated outcomes at hospital discharge (Aim 1b) and at 3-month follow-up (secondary outcomes; Aim 2). Experimental Approach. Pilot randomized controlled trial with blinded outcome assessment and 3-month phone-based follow-up.

Significance of the results. ARF patients experience significant anxiety during ICU stay, reporting feelings of terror, fear of death, and loss of control. Up to 50% of ARF patients report clinically significant anxiety at ICU discharge, and up to 40% report persistent symptoms up to 5 years after ICU. This project provides an essential foundation for evaluating a novel intervention, with a strong evidence-base outside of the ICU, to reduce anxiety in acute respiratory failure patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* English speaking and not aphasic
* ARF with mechanical ventilation via endotracheal tube > 24 hours
* Expected hospital stay of >7 days at time of eligibility
* Alert (ie, Richmond Agitation Sedation Scale sedation score = -1, 0, or 1)
* Not delirious (ie, negative Confusion Assessment Method -ICU score)
* Presence of anxiety symptoms (Visual Analog Scale-Anxiety score ≥50)**

Exclusion Criteria:

* Pre-existing cognitive impairment (AD-8 score ≥2)
* History of major psychiatric illness (i.e., psychotic disorder, bi-polar disorder, suicide attempt in past 24 months, pervasive developmental disorder, active substance use disorder)
* Declines or incapable of informed consent
* Anticipated discharge to hospice, primary focus on palliative care, or >90% probability of in-hospital death

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Satisfaction Questionnaire | 5 weeks post-enrollment
  Treatment Satisfaction Questionnaire (TSQ) ranges from 0-21, with higher scores representing greater satisfaction. Items (e.g., "useful", "liked it," "perceived symptom improvement") are scored based on a Likert scale, ranging from 0= "not at all" to 7= "very much so." Higher scores indicate higher satisfaction
average accrual rate of 2 patients/month across all patients | 3 years
  treatment feasibility objective
treatment feasibility as assessed by sessions completed | 5 weeks post enrollment
  treatment feasibility as assessed by >70% of intervention sessions completed
treatment feasibility as assessed by drop out rate | 3 years
  treatment feasibility as assessed by <15% drop-out across intervention arm

SECONDARY OUTCOMES:
Visual Analog Scale - Anxiety | at hospital discharge (up to 12 weeks after randomization), 5 weeks post enrollment, 3 months
  the 100 mm Visual Analog Scale for Anxiety (VAS-A.) Scores range from "not anxious at all" (0 mm) to "the most anxious I have ever felt" (100 mm).
State Anxiety Inventory | at hospital discharge (up to 12 weeks after randomization), immediately post intervention, 5 weeks post intervention, 3 months
  The State Anxiety Inventory (SAI) is a 6 -item, abbreviated version of the original State Trait Anxiety Inventory, validated in ARF patients. The SAI assesses current emotional state using a Likert scale ranging from 1 "not at all" to 4 "very much," has a range of 0-24, and has been validated in ARF patients in the ICU. Higher score, higher anxiety.
Hopkins Rehab Engagement Scale | at hospital discharge (up to 12 weeks after randomization)
  The Hopkins Rehabilitation Engagement Scale 5-item scale for use in rating behavioral observations of patients during acute inpatient rehabilitation. Score ranges from 5 to 30 with higher scores representing better rehabilitation engagement.
Self Efficacy for Managing Chronic Disease Rating Scale | at hospital discharge (up to 12 weeks after randomization), 3 month followup
  The Self-Efficacy to Manage Chronic Disease Scale is made up of 6-items on a visual analog scale, ranging from 1 (not at all confident) to 10 (totally confident). Total scores range from 10-60. Higher scores represent greater confidence to manage chronic disease.
Hospital Anxiety and Depression Scale | at hospital discharge (up to 12 weeks after randomization), 3 month followup
  Hospital Anxiety and Depression Scale (HADS)is a 14-item measure with a likert response scale 0 "not at all" to 3 (stem varies). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). Higher scores suggest higher depression or anxiety symptoms.
Quality of Life as assessed by the European Quality of Life Scale (EQ-5D) | 3 month follow up
  European Quality of Life Scale, part of the NHLBI Core Outcome Measure Set for ARF survivors.
  The EQ-5D is a 6-item health-related quality of life measure recommended for use with ICU survivors. It provides utility estimates with US norms. Index scores range from -0.59 to 1, where 1 suggests better health state.
Post Traumatic Stress Disorder as assessed by the Impact of Events Scale - 6 | 3 month follow up
  Impact of Event Scale - 6 item (IES-6) is a post-traumatic stress disorder symptom measure, part of the NHLBI Core Outcome Measure Set for ARF survivors. Higher scores indicate more PTSD symptoms. Score range is 0-24.
Healthcare Utilization as assessed by Healthcare Utilization interview | 3 month follow-up
  The Healthcare Utilization Survey (HUS) is a structured interview assessing hospitalizations, nursing facility stays, rehabilitation facility stays, as well as number and type of outpatient provider visits.
Montreal Cognitive Assessment - Blind | 3 month follow up
  cognitive screen, part of the NHLBI Core Outcome Measure Set for ARF survivors
  The Montreal Cognitive Assessment - Blind (MOCA) is a 13-item cognitive screening instrument. Higher scores are better. Possible range = 0- 30

CONTACTS AND LOCATIONS:
Overall Officials: Megan Hosey, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] May AD, Parker AM, Caldwell ES, Hough CL, Jutte JE, Gonzalez MS, Needham DM, Hosey MM. Provider-Documented Anxiety in the ICU: Prevalence, Risk Factors, and Associated Patient Outcomes. J Intensive Care Med. 2021 Dec;36(12):1424-1430. doi: 10.1177/0885066620956564. Epub 2020 Oct 9. PMID 33034254
- [Background] Hosey MM, Wegener ST, Hinkle C, Needham DM. A Cognitive Behavioral Therapy-Informed Self-Management Program for Acute Respiratory Failure Survivors: A Feasibility Study. J Clin Med. 2021 Feb 20;10(4):872. doi: 10.3390/jcm10040872. PMID 33672672
- [Background] Chlan L, Savik K. Patterns of anxiety in critically ill patients receiving mechanical ventilatory support. Nurs Res. 2011 May-Jun;60(3 Suppl):S50-7. doi: 10.1097/NNR.0b013e318216009c. PMID 21543962